CLINICAL TRIAL: NCT02512146
Title: The Expression of the Ionotropic Glutamate Receptors in Colon of IBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2015SDU-QILU-G03
Record Dates: First submitted 2015-07-19; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Ionotropic glutamate receptors
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Taken biopsies during Colonoscopy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Irritable bowel syndrome: Patients meeting Rome III criteria of irritable bowel syndrome. Intervention: colonoscopy.
  Interventions: Procedure: colonoscopy
- Normal controls: Asymptomatic individuals for health surveillance or patients for follow up after polypectomy.
  Intervention: colonoscopy.
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — Patients will undergo colonoscopy and participants will get biopsies from the colon.

SUMMARY:
The study aims to determine the expression of the ionotropic glutamate receptors in colon of irritable bowel syndrome (IBS) patients and evaluate the relationship between the ionotropic glutamate receptors and IBS symptoms.

DETAILED DESCRIPTION:
Ionotropic glutamate receptors participate in pain in nervous system. In this study,participants will examine the expression of the ionotropic glutamate receptors in colon of irritable bowel syndrome (IBS) patients and evaluate the relationship between the ionotropic glutamate receptors and IBS symptoms.

Participants may futher study the mechanism using cell experiment.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting IBS Rome III criteria. Asymptomatic individuals for health surveillance or patients for follow up after polypectomy.

Exclusion Criteria:

Patients with known cancers or abdominal surgery. Alarm symptoms such as anaemia, gastrointestinal bleeding or obstruction, marked weight loss, abdominal mass. Patients who are unwilling to sign or give the informed consent form. Patients with impaired cardiac, liver or renal function. Patients with coagulopathy. Patients with pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients underwent colonoscopy in Qilu Hospital outpatient and inpatient department.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
the expression of the ionotropic glutamate receptors | 4 months
  Participants will examine the expression level of ionotropic glutamate receptors using quantitative real-time RT-PCR and western blot ,examine the distribution using immunohistochemy.
the relationship between the ionotropic glutamate receptors and IBS symptom | 6 months
  Symptoms will be assessed though the severity of abdominal pain or discomfort and seizure frequency.Participants will evaluate the relationship between the expression level or the distribution of ionotropic glutamate receptors and IBS symptom. If there is a link between them, participants will study the underlying molecular mechanisms.

CONTACTS AND LOCATIONS:
Overall Officials: xiuli zuo, PHD, Study Director — Department of Gastroenterology, Qilu Hospital
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China